CLINICAL TRIAL: NCT06613048
Title: Effect of Breathing Exercises Applied to Hemodialysis Patients on Anxiety, Fatigue and Quality of Life
Acronym: Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amasya University (Other)
Responsible Party: Principal Investigator, Mahmut Zengin, Director, Amasya University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: AmasyaU-MZ-673
Record Dates: First submitted 2024-09-22; First posted 2024-09-25 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Exercise; Hemodialysis
Keywords: Anxiety; Fatigue; quality of life
MeSH Terms: conditions — Motor Activity; Anxiety Disorders; Fatigue | interventions — Breathing Exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (breathing exercise) (Experimental): The researcher has a certificate in breathing exercises. Those who consent to participate in the study that meets the research criteria will be given training with a prepared training brochure about correct breathing technique, introduction and function of the diaphragm muscle, box breathing technique, diaphragm breathing technique and benefits of correct breathing before the exercise.
  Box breathing technique will be applied in addition to standard treatment, 3 sets per day (morning, noon and evening) for 6 weeks, 10 repetitions in each set.
  Diaphragm breathing exercise will be applied in addition to standard treatment, lasting 2 minutes in the first week, then increasing each week and reaching 12 minutes in the 6th week, as 3 sets (morning, noon and evening).
  Interventions: Other: Breathing exercise
- Control (No Intervention): The control group will receive standard care. No intervention will be applied to these patients during the follow-up period, only data collection forms will be applied. Data collection forms will be collected in the same time period as the intervention group.

INTERVENTIONS:
Other: Breathing exercise — The researcher has a certificate in breathing exercises. Those who consent to participate in the study that meets the research criteria will be given training with a prepared training brochure about correct breathing technique, introduction and function of the diaphragm muscle, box breathing technique, diaphragm breathing technique and benefits of correct breathing before the exercise.
  Box breathing technique will be applied in addition to standard treatment, 3 sets per day (morning, noon and evening) for 6 weeks, 10 repetitions in each set.
  Diaphragm breathing exercise will be applied in addition to standard treatment, lasting 2 minutes in the first week, then increasing each week and reaching 12 minutes in the 6th week, as 3 sets (morning, noon and evening).
  Arms: Experimental (breathing exercise)

SUMMARY:
Breathing exercises are one of the non-pharmacological methods frequently used in health care in recent years. The aim of this study is to evaluate the effect of breathing exercises on fatigue, anxiety symptoms and quality of life in hemodialysis patients.

DETAILED DESCRIPTION:
Introduction: Breathing exercises are one of the non-pharmacological methods frequently used in health care in recent years.

Objective: The aim of this study is to evaluate the effect of breathing exercises on fatigue, anxiety symptoms and quality of life in hemodialysis patients.

Method: This study will be conducted using a randomized controlled experimental research design at the pre-test-post-test level. The research sample will consist of 58 hemodialysis patients who meet the inclusion criteria of the sample and who apply to the hemodialysis unit of a training and research hospital. The research data will be collected using the personal information form, Beck anxiety inventory, Piper fatigue scale and SF-12 quality of life scales. The pre-test data of the research will be filled in the first interview with the patients and the post-test data will be applied at the end of the 6th week.

Conclusion: Maintaining physical and psychological comfort and improving the quality of life of patients receiving hemodialysis treatment are among the primary responsibilities of the nurse. In this regard, it is predicted that breathing exercises will be beneficial in controlling physical and psychological symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Being over the age of 18
* Being willing to participate in the study
* Speaking and understanding Turkish
* Having started hemodialysis treatment at least 6 months ago

Exclusion Criteria:

* Being on hemodialysis treatment with a diagnosis of stage 4 renal failure
* Being on hemodialysis treatment due to acute renal failure
* Having a malignancy related to the respiratory system (bronchus or lung)
* Having chest pain

  . -Having previously done box breathing and diaphragmatic breathing exercises/receiving training
* Having cognitive dysfunction
* Not giving consent to participate in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2025-02-17 (Actual); Primary Completion 2025-05-26 (Actual); Study Completion 2025-06-23 (Actual)

PRIMARY OUTCOMES:
Beck Anxiety Inventory | 6 week
  Beck Anxiety Inventory (BAI) is designed to measure the frequency of anxiety symptoms experienced by an individual. The scale, consisting of 21 items, is a Likert-type assessment scale scored between 0-3. Individuals rate each item by giving a score between 0-3 to determine how uncomfortable they have felt for the symptom in each item "including the day of the application, in the last week". The scale scores between 0-63. The high total score indicates the high level of anxiety experienced by the person. While 13 of the items describe physical symptoms, 3 reveal the cognitive aspects of anxiety. 3 items have a physical quality as well as a cognitive quality. Therefore, the BAI includes physiological, affective and cognitive symptoms of anxiety. The Cronbach Alpha value of the scale was determined as 0.92.
Quality of Life Scale | 6 week
  Quality of Life Scale (SF-12): SF-12; consists of two dimensions measuring physical (6 statements) and mental/psychological (6 statements) functioning. It includes various Likert-type statements (2-point Likert; yes-no or 5-point Likert; always, often, sometimes, very little, never etc.) regarding general health status, activity limits, depression, energy level etc. High scores indicate high quality of life.
Piper Fatigue Scale | 6 week
  Piper Fatigue Scale (PFS): PFS consists of 22 questions and subjectively evaluates fatigue perception. It has four sub-dimensions: the behavior/severity sub-dimension, which evaluates the effect and severity of fatigue on daily life activities; the affective sub-dimension, which covers the emotional meaning attributed to fatigue; the sensory sub-dimension, which reflects the mental, physical and emotional symptoms of fatigue; and the cognitive/spiritual sub-dimension, which reflects the degree to which fatigue affects cognitive functions and mood. The total score of the scale varies between 0 and 10. A score of 0 indicates no fatigue, 1-3 indicates mild fatigue, 4-6 indicates moderate fatigue, and 7-10 indicates severe fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Mahmut Zengin, Study Chair — Amasya University
Locations (1):
- Neşe Uysal, Amasya, Turkey (Türkiye)